CLINICAL TRIAL: NCT03545178
Title: Systematic Evaluation of Continuous Glucose Monitoring Data to for the Development of Clinical Solutions
Brief Title: Systematic Evaluation of Continuous Glucose Monitoring Data
Acronym: SECOND
Status: Completed | Type: Observational
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Other Study IDs: 2018-00207
Record Dates: First submitted 2018-04-18; First posted 2018-06-04 (Actual); Last update posted 2019-08-13 (Actual); Status verified 2019-08

CONDITIONS: Diabetes Mellitus
Keywords: white coat adherence; continuous glucose monitoring; flash glucose monitoring; hypoglycemia prediction; deep learning algorithm
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Diabetic patients using CGM/FGM: Evaluation of glucose control and application of hypoglycemia prediction models in diabetic patients wearing CGM and/or FGM devices for at least 50% of the time during the last 4 weeks prior to the medical consultation.
  Interventions: Behavioral: glucose control (Substudy A); Diagnostic Test: hypoglycemia prediction (Substudy B)

INTERVENTIONS:
Behavioral: glucose control (Substudy A) — Comparison of glucose values during days 0 - 3 with days 4 - 28 and 0 - 7 with days 8 - 28 before a medical consultation at the diabetes clinic in patients suffering from diabetes and wearing a continuous glucose monitoring and/or flash glucose monitoring device
Diagnostic Test: hypoglycemia prediction (Substudy B) — Use of CGM/FGM data to develop and evaluate a neural network based hypoglycemia prediction model

SUMMARY:
This study retrospectively evaluates continuous glucose monitoring (CGM) and flash glucose monitoring (FGM) data and pursues two main objectives: First, the investigators analyze if glucose values are better controlled in the days directly before a consultation at our tertiary referral centre (so called "white coat adherence"). Second, the investigators use the collected CGM and FGM data to develop a hypoglycemia prediction model.

DETAILED DESCRIPTION:
Substudy A.) Presence of white coat adherence in diabetic patients:

The investigators aim at evaluating the existence of a so called "white coat adherence" with regard to diabetes control, which means that blood-glucose is better controlled in the days immediately prior to a consultation at the diabetes clinic compared to the time-period further back. To analyse this phenomenon, the investigators use continuous glucose monitoring (CGM) and flash glucose monitoring (FGM) of diabetic patients and compare CGM-/FGM data of the last three days prior to the consultation with the CGM-/FGM data of the days 4-28 prior to the consultation, as well as the last seven days prior to the consultation with days 8-28 prior to the consultation.

Substudy B.) Retrospective data collection for the development and evaluation of a hypoglycemia prediction model:

Scope of the study is to use retrospective data for training and evaluation of a deep recurrent neural network based system for predicting the onset of hypoglycemic event at least 20 min ahead in time. The study aims to: I, assess the ability of deep learning algorithm to predict hypoglycemic events using the data collected during substudy 1. II, assess the ability of global model to be personalized using the data collected during sub-study 1. III, investigate the amount of "history" to be involved to achieve maximum performance in terms of prediction ability. IV, develop a global model, which can be easily further personalized to achieve optimum prediction performance per patient.

ELIGIBILITY:
Inclusion Criteria:

* Diabetes mellitus
* CGM and/or FGM available for at least 50% of the time in last 4 weeks before consultation
* Written informed general consent for the retrospective analysis of data

Exclusion Criteria:

* Pregnancy

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients suffering from diabetes mellitus controlled at our tertiary referral centre using a CGM/FMG device for at least 50% of the time
Sampling Method: Non-Probability Sample
Enrollment: 384 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2019-07-19 (Actual); Study Completion 2019-07-19 (Actual)

PRIMARY OUTCOMES:
Change of time in target glucose range day 0-3 compared to day 4-28 and day 0-7 compared to day 8-28 prior to consultation (for Substudy A) | 01.01.2013 - 31.07.2018; outcome assessed at study end
  The time spent in the target glucose range from 3.9 to 10.0 mmol/l assessed by CGM/FGM.
Hypoglycemia prediction (for Substudy B) | 01.01.2013 - 31.07.2018; outcome assessed at study end
  Proportion of times a deep learning based algorithm can predict a hypoglycemic event (BG <4.0 mmol/l) at least 20 min ahead in time?

SECONDARY OUTCOMES:
Change of time above and below glucose target range day 0-3 compared to day 4-28 and day 0-7 compared to day 8-28 prior to consultation (for Substudy A) | 01.01.2013 - 31.07.2018; outcome assessed at study end
  The time spent above and below the target glucose (3.9 to 10.0 mmol/l) assessed by CGM/FGM.
Change of average and standard deviation glucose day 0-3 compared to day 4-28 and day 0-7 compared to day 8-28 prior to consultation (for Substudy A) | 01.01.2013 - 31.07.2018; outcome assessed at study end
  Average and standard deviation glucose levels based on CGM/FGM data
Sensor wearing time day 0-3 compared to day 4-28 and day 0-7 compared to day 8-28 prior to consultation (for Substudy A) | 01.01.2013 - 31.07.2018; outcome assessed at study end
  Time CGM-/FGM sensor has been worn (%)
Change of coefficient of variation (CV) day 0-3 compared to day 4-28 and day 0-7 compared to day 8-28 prior to consultation (for Substudy A) | 01.01.2013 - 31.07.2018; outcome assessed at study end
  Coefficient of variation (CV) based on CGM/FGM data
Change of time in hypoglycemia day 0-3 compared to day 4-28 and day 0-7 compared to day 8-28 prior to consultation (for Substudy A) | 01.01.2013 - 31.07.2018; outcome assessed at study end
  The time with glucose levels < 3.0 based on CGM/FGM data
Change of time in hyperglycemia day 0-3 compared to day 4-28 and day 0-7 compared to day 8-28 prior to consultation (for Substudy A) | 01.01.2013 - 31.07.2018; outcome assessed at study end
  The time with glucose levels in the significant hyperglycaemia, as based on CGM/FGM (glucose levels > 13.9 mmol/l)
Change of mean amplitude of glucose excursion (MAGE) day 0-3 compared to day 4-28 and day 0-7 compared to day 8-28 prior to consultation (for Substudy A) | 01.01.2013 - 31.07.2018; outcome assessed at study end
  The mean amplitude of glucose excursion assessed by CGM/FGM

OTHER OUTCOMES:
Change of total, basal and bolus insulin dose day 0-7 compared to day 8-28 prior to consultation (for Substudy A) | 01.01.2013 - 31.07.2018; outcome assessed at study end
  Total, basal and bolus insulin dose based on data of continuous subcutaneous insulin infusion data in patients treated with insulin pumps
Change of periods with glucose below 3.0mmol/l for at least 15 minutes day 0-3 compared to day 4-28 and day 0-7 compared to day 8-28 prior to consultation (for Substudy A) | 01.01.2013 - 31.07.2018; outcome assessed at study end
  Duration of periods when sensor glucose values was below 3.0mmol/l for at least 15 minutes
Change of periods with glucose above 13.9mmol/l for at least 15 minutes day 0-3 compared to day 4-28 and day 0-7 compared to day 8-28 prior to consultation (for Substudy A) | 01.01.2013 - 31.07.2018; outcome assessed at study end
  Duration of periods when sensor glucose values was above 13.9mmol/l for at least 15 minutes
Change of mean of daily differences (MODD) day 0-3 compared to day 4-28 and day 0-7 compared to day 8-28 prior to consultation (for Substudy A) | 01.01.2013 - 31.07.2018; outcome assessed at study end
  Mean of daily differences (MODD) based on CGM/FGM data

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Zueger, MD, Principal Investigator — Department of Diabetes, Endocrinology, Clinical Nutrition and Metabolism, Inselspital, Bern University Hospital, University of Bern, 3010 Bern, Switzerland; Christoph Stettler, Prof., Study Director — Department of Diabetes, Endocrinology, Clinical Nutrition and Metabolism, Inselspital, Bern University Hospital, University of Bern, 3010 Bern, Switzerland
Locations (1):
- Inselspital, Bern University Hospital, University of Bern, Bern, Canton of Bern, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided